CLINICAL TRIAL: NCT02832609
Title: Mechanisms of Orthopnea in Stable Obese Patients
Acronym: OBAIRWAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009-574
Record Dates: First submitted 2016-07-07; First posted 2016-07-14 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2016-07

CONDITIONS: Obesity
Keywords: closing volume; expiratory flow limitation; obesity; orthopnea
MeSH Terms: conditions — Obesity; Dyspnea | interventions — Supine Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- sitting position (No Intervention): measurement in the sitting position
- supine position (Active Comparator): measurement in the sitting position
  Interventions: Other: Supine

INTERVENTIONS:
Other: Supine — measurements after 30 minutes in complete supine position
  Arms: supine position

SUMMARY:
The purpose of this study is to study the role of closing volume as a determinant of orthopnea in stable obese subjects. The investigators hypothesized that: (1) increase in closing volume in supine position would be greater in orthopneic than in non-orthopneic subjects, and (2) the relationship of change in closing volume to change in dyspnea with position would be dependent on expiratory flow limitation in the sitting position.

In stable obese subjects, in sitting and supine positions, the investigators measured Borg dyspnea score, static lung volumes, expiratory flow limitation, and single-breath nitrogen expiration test, from which the investigators determined closing volume and closing capacity, slope of phase III, and opening capacity.

Orthopnea was defined as any increase in the Borg score in the supine position from its value in the sitting position

ELIGIBILITY:
Inclusion Criteria:

* obese (BMI ≥ 30)
* stable condition
* 20 < Age < 60 years

Exclusion Criteria:

* other respiratory disorder (COPD)
* left cardiac insufficiency

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
closing volume by nitrogen washout method | 30 minutes after changing position (hour 2)

SECONDARY OUTCOMES:
static lung volumes by plethysmography | 30 minutes after changing position (hour 2)
  static lung volumes are composed of vital capacity, FEV1, inspiratory capacity, and reserve expiratory volume and are measured by plethysmography
expiratory flow limitation by NEP test | 30 minutes after changing position (hour 2)
  NEP test

CONTACTS AND LOCATIONS:
Overall Officials: Claude Guérin, Prof, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices civils de lyon, Hôpital de la Croix-Rousse - Réanimation, Surveillance Continue Médicales et Assistance Respiratoire, Lyon, France

REFERENCES:
- [Result] Perino E, Nesme P, Germain M, Guerin C. Mechanisms of Orthopnea in Stable Obese Subjects. Respir Care. 2016 Aug;61(8):1015-22. doi: 10.4187/respcare.04146. Epub 2016 Apr 5. PMID 27048626